CLINICAL TRIAL: NCT04674371
Title: German Point Prevalence Study on Central Venous Catheter
Brief Title: German Point Prevalence Study on CVC
Status: Completed | Type: Observational
Sponsor: Wolfram Schummer, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Wolfram Schummer, MD, PhD, PD Dr. med. Dr. med. habil., Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin
Organization: Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin (Other)
Other Study IDs: DRKS00016855; U1111-1229-1554 (Registry Identifier: World Health Organization [WHO] Registry Network)
Record Dates: First submitted 2020-12-13; First posted 2020-12-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-05

CONDITIONS: Data Collection
Keywords: Central venous catheter; central venous line; Catheterization, Central Venous / access; Catheterization, Central Venous / methods; Catheterization, Central Venous / instrumentation; Catheterization, Central Venous / adverse effects; Placement of larger catheters; Insertion of CVCs; Complication of CVCs; CVC misplacement; Ultrasonography, Interventional / adverse effects; Ultrasonography, Interventional / instrumentation; Ultrasonography, Interventional / methods; Electroctrocardiography, Radiography, Echocardiographie/ TEE; Vascular Access Devices / standards; Vascular Access Devices / trends; Critical Illness / therapy; Humans; Adults, Adolescents
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: central venous catheter insertion — Every operator should perform the CVC Insertion Procedure according to his common clinical practice.

SUMMARY:
It has now been 90 years since Werner Forssmann developed the CVC. Nowadays CVCs play an integral role for critically ill patients.

Despite the high number of central venous access devices inserted annually, there are limited data on the incidence of the associated procedural complications, many of which carry substantial clinical risk. This point was highlighted in recently published Association of Anaesthetists of Great Britain and Ireland "Safe vascular access 2016" guidelines and "Clinical guidelines on central venous catheterisation" in 2014 of the Swedish Society of Anaesthesiology and Intensive Care Medicine.

This German point prevalence study should identify the number of central venous catheter insertions and the incidence of various and especially serious mechanical complications across multiple hospital sites within one day.

Secondary aims are to identify the availability of resources and infrastructure to facilitate safe central venous catheter insertion and management of potential complications.

As much hospital sites as possible should participate and identify all adult central venous catheter insertions, with subsequent review of any complications detected.

Additionally, resources while inserting the CVC should be specified such as ultrasound for assessment of ultrasound anatomy and/or ultrasound-guidance. Furthermore, assessment of the CVC tip should be studied whether done during CVC placement with

* ECG-guidance or by
* transthoracic/transesophageal ultrasound with the Microbubble test or more conventional post hoc with
* bedside chest X-ray Any mechanical complication should be documented untill day three post insertion. The background is to identify possible perforations due to initially unfavorable CVC tip positions (angle > 40 ° to wall of the superior vena cava).

Participation in the study is open to all disciplines (anesthesia, intensive care, internal medicine, surgery, etc.) that regularly perform CVCs.

DETAILED DESCRIPTION:
Questions

* How experienced are the CVC operators?
* What are the demographics of the patients included?
* How many emergency patients will be included in the study?
* How is the distribution of the punctured vessels and that of the respective sides?
* How many puncture attempts are necessary to achieve a successful CVC placement and how often do problems with the Seldinger-wire occur?
* How often is ultrasound used to place a CVC and if so,

  1. Only for Screening?
  2. Puncture under ultrasound view?
* What is the distribution between short and long axis view?
* What catheter types and which caliber in French are being inserted?
* Catheter position control:

  1. by EKG-lead on Pmax or Pmax - x cm (withdroth)
  2. by means of transthoracic ultrasound and agitated NaCl solution
  3. by means of transesophageal echocardiography and NaCl solution
  4. by means of X-ray image
  5. other or missing position control
* Statement on the position of the CVC tip
* How common are CVC-malpositions and what is their distribution?
* Which complications occur within 72 h? Which measures do you require and how do they affect the respective patient?

ELIGIBILITY:
Age

* Inclusion criteria:

  * Adults
  * Young Adults
  * Children
  * Infants
  * Neonates
* Exclusion criteria:

  * None

Procedures

* Inclusion criteria:

  * Elective central venous access procedures
  * Emergency central venous access procedures
* Exclusion criteria:

  * None

Providers

* Inclusion criteria:

  * Anesthesiologists
  * Internist
  * Neurologist
  * Surgeon
  * Etc.
* Exclusion criteria:

  * None

Selection of catheter insertion site

* External jugular
* Internal jugular
* Subclavian
* Femoral

Complications

* Inclusion criteria:

  * Arterial cannulation/injury/cerebral embolization/hemorrhage
  * Catheter or wire shearing or loss
  * Lacerations of great vessels
  * Exsanguination
  * Hemo/pneumothorax; peritoneal hemorrhage
  * Pneumothorax
  * Tamponade
  * Tracheal injury
  * Air embolism
  * Heart puncture (tamponade)
  * Hemothorax
  * Stroke
  * Mortality
  * Number of attempts at central line placement
  * Failed insertion attempts
  * Successful, nontraumatic procedure
  * Wire, needle, catheter issues
* Exclusion criteria:

  * Infections or other complications not associated with central venous catheterization
  * Mechanical injury or trauma not associated with central venous catheterization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Over 2000 patients in Germany
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Patients Demographics | 17.05.2022
  All patients with a CVC Insertion on May 17th. 2022 in participating Hospitals independent of sex, age or BMI in kg/m^2 are eligible
Complications and malpositions | 17.05.2022-20.05.2022
  Which complications and malpositions occur within 72 h

SECONDARY OUTCOMES:
Percentage of the emergency procedure | 17.05.2022
  How many emergency patients will be included in the study
Distribution of the vessel sites und sides | 17.05.2022
  distribution of the punctured vessels (external jugular, internal jugular, subclavian, femoral
  ) and that of the respective sides
Experience of the operator | 17.05.2022
  Resident physician/ Specialist doctor
Puncture attempts | 17.05.2022
  How many puncture attempts are necessary to achieve a successful CVC
Type and caliber of catheter | 17.05.2022
  What catheter types and which caliber in French are being inserted
Wire problems/issues | 17.05.2022
  witch and how often do problems with the Seldinger-wire occur
Ultrasound assistance | 17.05.2022
  Screening / Online guidance / Short or long axis view
CVC tip position | 17.05.2022
  measures to ensure central venous catheter tip position (i.e. CXR, ECG method and ultrasound)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Schummer, MD, PhD, Study Chair — Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin
Locations (1):
- Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin e.V., Mitte, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt GA, Blaivas M, Conrad SA, Corradi F, Koenig S, Lamperti M, Saugel B, Schummer W, Slama M. Ultrasound-guided vascular access in critical illness. Intensive Care Med. 2019 Apr;45(4):434-446. doi: 10.1007/s00134-019-05564-7. Epub 2019 Feb 18. PMID 30778648
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Schummer W, Sakka SG, Huttemann E, Reinhart K, Schummer C. [Ultrasound guidance for placement control of central venous catheterization. Survey of 802 anesthesia departments for 2007 in Germany]. Anaesthesist. 2009 Jul;58(7):677-85. doi: 10.1007/s00101-009-1569-1. German. PMID 19547936
- [Background] Frykholm P, Pikwer A, Hammarskjold F, Larsson AT, Lindgren S, Lindwall R, Taxbro K, Oberg F, Acosta S, Akeson J. Clinical guidelines on central venous catheterisation. Swedish Society of Anaesthesiology and Intensive Care Medicine. Acta Anaesthesiol Scand. 2014 May;58(5):508-24. doi: 10.1111/aas.12295. Epub 2014 Mar 5. PMID 24593804
- [Background] Coe AJ. AAGBI Safe vascular access guidelines I. Anaesthesia. 2016 Aug;71(8):985. doi: 10.1111/anae.13553. No abstract available. PMID 27396261
- [Background] Bierman S. AAGBI safe vascular access guidelines II. Anaesthesia. 2016 Aug;71(8):985-6. doi: 10.1111/anae.13554. No abstract available. PMID 27396262
- [Background] Lathey RK, Jackson RE, Bodenham A, Harper D, Patle V; Anaesthetic Audit and Research Matrix of Yorkshire (AARMY). A multicentre snapshot study of the incidence of serious procedural complications secondary to central venous catheterisation. Anaesthesia. 2017 Mar;72(3):328-334. doi: 10.1111/anae.13774. Epub 2016 Dec 16. PMID 27981565

DOCUMENTS (1):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04674371/Prot_000.pdf